CLINICAL TRIAL: NCT03760315
Title: Department of Critical Care Medicine, Nanjing Zhong-Da Hospital, Southeast University School of Medicine,China;
Brief Title: mNGS vs Culture Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Ling Liu, Director, Southeast University, China
Other Study IDs: 20181127
Record Dates: First submitted 2018-11-28; First posted 2018-11-30 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Sepsis
Keywords: next- generation sequencing； blood culture；IDSeqTM Ultra
MeSH Terms: conditions — Sepsis | interventions — Blood Culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis: All enrolled patients
  Interventions: Diagnostic Test: blood mNGS (IDSeqTM Ultra); blood Culture

INTERVENTIONS:
Diagnostic Test: blood mNGS (IDSeqTM Ultra); blood Culture — take blood samples for mNGS and Culture at the same time in sepsis patients. No intervention on the treatment of the patients.

SUMMARY:
mNGS is popular in research and recently it has been used clinically to detect microbes in the blood or other secretion in infected patients for quicker ,broad and accurate detection of microbes. In ICU ,patients are critically ill and need quicker and accurate antibiotics use to stop the pathologic process. The purpose of this study was to determine whether the positive detection rate of pathogens in patients with sepsis by metagenomic full-targeted detection technology was higher than that in blood culture, and to determine whether the pathogens found in patients with sepsis by metagenomic full-targeted detection technology were important for clinical development. Anti-infective regimens can help.

DETAILED DESCRIPTION:
Sepsis patients in ICU were took blood culture sample and blood sample for mNGS test (IDSeqTM Ultra, Combing with Metagenomics and Pathogen/AMR/VF Probe Enrichment). Clinicians use their knowledge and experience to decide antibiotics use with the guide of Culture results or mNGS results. Validation with digital droplet PCR assays when metagenomic full-targeted assays identify pathogens not identified in conventional blood cultures The difference between the positive rate of mNGS and the positive rate of blood culture were recorded. Patient were followed at least 28 days after enrollment or an outcome indicator. Possible scenarios for detecting clinical impact were detected. Etiology, biochemical indicators, immune function, infection indicator, secondary infection, SOFA score and length of stay，outcome were recorded.

ELIGIBILITY:
Inclusion Criteria:

Age > 18years admit to ICU Meet the Sepsis 3.0 diagnostic criteria and suspected bloodstream infection, and the diagnosis of Sepsis ≤ 24 hours; Estimated ICU stay ≥ 24 hours; Informed consent;

Exclusion Criteria:

Severe organ dysfunction, expected death within 72 hours; Receive palliative care; Refuse to participate;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with sepsis and suspected bloodstream infection
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
difference of positive rate between mNGS and Culture | 28 day
  The difference between the positive rate of mNGS and the positive rate of blood culture.

SECONDARY OUTCOMES:
The difference between the positive rate of metagenomic full capture technology and the Category of Clinical Impact | 28 day
  Positive, Negative，None and Indeterminate
Change of SOFA | 7 day
  change of SOFA score (include each organ) at baseline, day 3 and day 7 clinical improvement :Improvement in 2 or more clinical signs and symptoms no requirement for additional antibacterial treatment Clinical failure:Persistence or progression of baseline signs and symptoms
Mortality | During hospitalization
  28 day，ICU and hospital mortality Documented microbiologic eradication:Absence of primary microbe from infection site Presumed microbiologic eradication:Clinical cure without available microbiologic culture data Presumed microbiologic persistence:Clinical failure in the absence of any microbiologic data Documented microbiologic persistence:Continued presence of MRSA based on microbiologic culture Superinfection: Clinical failure and isolation of a pathogen not present at baseline at the original infection site
Length of stay | During hospitalization
  ICU and hospital length of stay
Anti-infective treatment adjustment | 28 day
  each Anti-infective treatment adjustment

OTHER OUTCOMES:
pathogen | 28 day
  all the detect pathogens from mNGS and blood culture
secondary infection | 28 day
  infection secondary to the primary infection

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, MD, Study Director — Southeast University, China
Locations (1):
- Nanjing Zhong-Da Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Sun Q, Teng R, Shi Q, Liu Y, Cai X, Yang B, Cao Q, Shu C, Mei X, Zeng W, Hu B, Zhang J, Qiu H, Liu L. Clinical implement of Probe-Capture Metagenomics in sepsis patients: A multicentre and prospective study. Clin Transl Med. 2025 Apr;15(4):e70297. doi: 10.1002/ctm2.70297. PMID 40181528